CLINICAL TRIAL: NCT00195013
Title: A Randomized Placebo-controlled Trial of Glutamine to Reduce the Signs and Symptoms of Peripheral Neuropathy in Breast Cancer Patients With a Mild Peripheral Neuropathy Receiving Paclitaxel Chemotherapy
Brief Title: Randomized Placebo-Controlled Trial of Glutamine for Breast Cancer Patients With Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0309006308
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Neuropathy; Breast Cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Glutamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): 10 grams three times a day (orally) for four days and then stop
  Interventions: Drug: glutamine
- Placebo (Placebo Comparator): 10 grams three times a day (orally) for four days and then stop
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: glutamine — 10 grams three times a day (orally) for four days and then stop
  Other Names: NutreStore
  Arms: Glutamine
Drug: Placebo — 10 grams three times a day (orally) for four days and then stop
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Patients with breast cancer receiving paclitaxel chemotherapy who have mild symptoms of peripheral neuropathy will receive glutamine or placebo to try and improve symptoms.

DETAILED DESCRIPTION:
1. Determine whether oral glutamine supplementation can reduce the symptoms and signs of peripheral neuropathy.
2. Determine whether alterations in the symptoms and signs of peripheral neuropathy are correlated with an alteration of circulating nerve growth factor or insulin-like growth factor levels.
3. Assess whether oral glutamine affects circulating nerve growth factor or insulin-like growth factor levels.
4. Assess whether glutamine interferes with paclitaxel pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed breast cancer, Stage I, II, III or IV or other solid tumors.
2. Patients must be receiving weekly paclitaxel or nab-paclitaxel chemotherapy or have recently completed paclitaxel or nab-paclitaxel chemotherapy and have at least a Grade I peripheral neuropathy (see Appendix A) because of therapy.
3. Because no dosing or adverse event data are currently available on the use of glutamine in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
4. ECOG performance status <1 (Karnofsky >90%).
5. Life expectancy of greater than 3 months.
6. Patients must have sufficient organ and marrow function so that paclitaxel treatment can be administered.
7. The effects of glutamine on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have experienced prior neuropathies not associated with chemotherapy
2. Patients may not be receiving any other investigational agents.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. There are no known allergies associated with glutamine.
5. Uncontrolled intercurrent illness that render the patient ineligible to receive paclitaxel chemotherapy.
6. Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with glutamine. Breastfeeding should also be discontinued if the mother is treated with glutamine.
7. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with glutamine. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
8. Concurrent chemotherapy with another drug known to cause neuropathy (CDDP or CBDCA or oxaliplatin) are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Vahdat, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glutamine | Placebo
Started | 14 | 16
Completed | 12 | 15
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glutamine | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 3 | 2 | 5
Age, Continuous [Median (Full Range); unit: years] | 58 [39 to 69] | 55 [37 to 74] | 58 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Peripheral Neuropathy Score
Description: Used the clinical total neuropathy score scale (TNSc). The presence of sensory, motor, pin sensibility, vibration sensibility, DTR, autonomic symptoms was assessed. For each item, the possible score ranged between 0 (normal) and 4 (worst possible result).
  Outcomes calculated as neuropathy score value at 10 Weeks minus neuropathy score value at Baseline. Increased score value indicates increased neuropathy severity.
Time Frame: Duration of study, approximately 10 weeks per subject
Measure: Mean (Full Range); unit: Change in Total Neuropathy Score
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 14 | 16
Change in Total Neuropathy Score | 0.3 [-5 to 3] | 0.9 [-6 to 7]

ADVERSE EVENTS:
Arm/Group | Glutamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes